CLINICAL TRIAL: NCT07278622
Title: Feasibility Testing and Process Evaluation of a Virtual Group Preoperative Prehabilitation Education Intervention (GoPREPARE)
Brief Title: Virtual Group Prehabilitation Education (Surgery School) Feasibility Trial
Acronym: GoPREPARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University Hospital Plymouth NHS Trust (Other); University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RHM CRI0467
Record Dates: First submitted 2025-08-06; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-07

CONDITIONS: Cancer Surgery; Elective Surgery; Patient Education; Prehabilitation
Keywords: surgery school; prehabilitation; patient education; perioperative care

STUDY DESIGN:
Intervention Model Description: Intervention versus standard care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GoPREPARE Education Intervention (Experimental): A 1.5 live education webinar delivered to groups of patients and their carers before surgery. Delivered by health care professionals.
  Interventions: Other: GoPREPARE
- Standard Care (No Intervention): Patients will be given a standard prehabilitation leaflet

INTERVENTIONS:
Other: GoPREPARE — GoPREPARE is a live interactive virtual education and behaviour change intervention delivered by healthcare professionals to groups of patients and their family, friends and carers which aims to prepare them for major cancer surgery.
  Arms: GoPREPARE Education Intervention

SUMMARY:
One in four patients requiring planned major surgery have complications. Prehabilitation; which involves increasing physical activity, improving nutrition and supporting emotional well-being prior to surgery can reduce these complications and improve recovery. Group preoperative prehabilitation classes (surgery schools) are advocated by the Centre for Perioperative Care and are standard care in many hospitals, despite a lack of evidence for their effectiveness in improving patient outcomes. In phase 1 an 2 of this research investigators used patient experiences and co-participatory methods to optimise an existing intervention to make it as acceptable and as engaging as possible. The resulting education package is called 'GoPREPARE'

Investigators now intend to test the practicalities of trialing GoPREPARE on preoperative patients with cancer. 24 patients awaiting surgery will be recruited from University Hospital Plymouth and randomly allocated equally to: Group - GoPREPARE and Group 2- standard care. Participants will complete lifestyle questionnaires before during and after their hospital stay. To evaluate the experience, ~8 participants will be interviewed. 5 clinical staff involved in the trial will also take part in a focus group. The information collected will be analysed to assess if it is feasible to conduct a larger trial.

DETAILED DESCRIPTION:
See uploaded protocol

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing elective surgery for any body cavity cancer with curative intent.
* Adults with more than 3 weeks before planned surgery
* Adults without previous experience of prehabilitation.

Exclusion Criteria:

* Children
* Adults who lack mental capacity.
* Adults who do not understand spoken English.
* Previous experience of prehabilitation.
* Previous surgery for cancer
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility Outcome Measure: Proportion of eligible patients recruited | From start of recruitment to recruitment closing. Approximately 6 months
  E.g. number recruited compared with number eligible.
Feasibility Outcome Measure: Number of patients who decline and reasons for decline | During recruitment period approximately 6 months
  Number of patients who decline to take part in the study and reasons.
Feasibility Outcome Measure: Number of missed eligible patients | From start of trial to recruitment closing. Approximately 6 months
  Number of eligible patients not approached and reasons.
Feasibility Outcome Measure: Number of patients who remain in the trial for the full duration | From recruitment through to three month post surgery follow up. (Approx 4 months total)
  Retention of participants to trial and follow up. E.g. number of patients who remain in the trial until the follow up completed.
Feasibility Outcome Measure: Participant experience of GoPREPARE | 2 months after surgery, approximately 3 months after enrollment
  Participant experience of GoPREPARE. Interviews will be undertaken and experience captured through qualitative thematic analysis.
Feasibility Outcome Measure: Staff experiences of taking part in GoPREPARE trial | At end of recruitment period. Approximately months 6-8
  Staff experiences of delivering GoPREPARE trial. A focus group will be conducted at the end of the trial and experiences captured through thematic qualitative analysis.

SECONDARY OUTCOMES:
Suitability and sensitivity of outcome measures: Return rate and completeness of questionnaires | From recruitment through to three month post surgery follow up. (Approx 4 months total)
  Return rate and completeness of questionnaires.
Suitability and sensitivity of outcome measures: Average time participants wear their accelerometer | From recruitment for two weeks, for one further week at around 3 months post surgery.
  Participant compliance with wearing accelerometer and usefulness of data collected.
Suitability and sensitivity of outcome measures: Adverse events | From recruitment through to three month post surgery follow up. (Approx 4 months total)
  Documentation of adverse events occurring during trial duration
Suitability and sensitivity of outcome measures: Number of days spent in hospital following surgery | In hospital stay approx 3-5 weeks following recruitment
  Date of hospital admission minus date of discharge would equal length of post-operative stay (LOS)
Suitability of sensitivity of outcome measurements: Incidence of postoperative morbidity/mortality | From discharge from hospital to three month follow up
  On day of discharge and at 3 month follow up patient's surgical complications (if any) will be graded using the Clavien-Dindo classification of surgical complications This classification is used to assess overall hospital morbidity following surgical procedures. Patients are graded as 0 (no complications) or Grade I-V based on the level of complication, including the number of organ system involvement. Grade V is defined as death of a patient. A record of the Comprehensive Complication Index (CCI) - an update of the Clavien-Dindo classification will also be collected.
Suitability and sensitivity of outcome measures: Post-operative recovery behaviour compliance | First three days after having had surgery
  Post-operative recovery behaviour compliance measured using a questionnaire to capture frequency of postoperative breathing exercises, and the restarting of eating, drinking and mobilising by day three post surgery questionnaire
Suitability and sensitivity of outcome measures: Physical Activity 1 | At baseline for two weeks and at three months post surgery
  Number of steps while active using a triaxial accelerometer eg. Actigraph
Suitability and Sensitivity of Outcome Measures: Physical Activity 2 | At baseline, prior to admission for surgery and at 3 months post surgery
  Godin Leisure Time and Exercise questionnaire - A self-reported measure of physical activity
Suitability and Sensitivity of Outcome Measures: Health Related Quality of Life | At baseline, prior to admission for surgery and at three month follow up post surgery.
  Changes in health related quality of life measurements using validated questionnaires; including:
  EQ-5D-5L is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status that can be used in the clinical and economic evaluation of health care as well as in population health surveys
Suitability and Sensitivity of Outcome Measures: Nutrition 1 | At baseline, before admission to hospital for surgery and at three month follow up post surgery
  Height (cms) and weight (kg) will be combined to report BMI in kg/m^2
Suitability and Sensitivity of Outcome Measures: Nutrition 2 | At baseline, prior to admission for surgery and at three month follow up post surgery
  Patient self-completing Worldwide Cancer Research (WCRF) Screening and food frequency questionnaire. This asks about things like diet, processed foods, meat, drinks, answers can then be used to score how closely the lifestyle follows WCRF's cancer-prevention recommendations.
Suitability and Sensitivity of Outcome Measures: Mental Well-being | At baseline, before admission to hospital for surgery and at three month follow up post surgery
  Anxiety and depression will be measured using the Hospital Anxiety and Depression Scale (HADS)
  A tick box questionnaire relating to anxieties and depression that a patient might have felt over the past week. Choices are most of the time, a lot of the time, from time to time, and not at all for most questions.
Suitability and Sensitivity of Outcomes Measures: Smoking | At baseline, preadmission for surgery and three months follow-up post surgery.
  Smoking habits measured using GATS (Global Adult Tobacco Survey) It asks about smoking and smokeless tobacco use, quitting habits and exposure to secondhand smoke.
Suitability and sensitivity of outcome measure: Alcohol Intake | At baseline, preadmission for surgery and at three month follow-up post surgery.
  Alcohol intake to be measured using the AUDIT-C is a short alcohol screening test used to check whether someone's drinking might be risky or harmful.

CONTACTS AND LOCATIONS:
Overall Officials: Denny Z Levett, PhD, Study Director — Universal Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospitals Plymouth NHS Trust, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data including demographics or participants and direct quotes following the process evaluation interviews will be shared in academic journals. All data will be anonymised.